CLINICAL TRIAL: NCT07231835
Title: RECORD-DCB: Registry of Coronary Disease Outcomes Revascularizing With Drug-Coated Balloons
Brief Title: Registry of Coronary Disease Outcomes Revascularizing With Drug-Coated Balloons
Acronym: RECORD-DCB
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Bimmer Claessen, md phd, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2025.0981
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Percutaneous Coronary Intervention (PCI); Drug Coated Balloon; Paclitaxel; CAD - Coronary Artery Disease; ACS (Acute Coronary Syndrome); Stable Coronary Artery Disease (CAD), Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this registry is to systematically collect and analyze real-world data on all patients undergoing PCI with the Protégé paclitaxel-eluting DCB to evaluate procedural outcomes, long-term efficacy, and safety across various clinical indications. This registry aims to assess the clinical effectiveness of DCB therapy across diverse patient populations, including those with stable coronary artery disease (CAD) and acute coronary syndromes (ACS), as well as various lesion subsets, encompassing (but not limited to) in-stent restenosis (ISR), de novo coronary lesions, small vessel disease, bifurcation and calcified lesions, coronary bypass graft lesions, and patients at high risk of bleeding. Additionally, the study aims to identify predictors of success, complications, and optimal treatment strategies to further refine the use of DCBs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PCI with the Protégé paclitaxel-eluting DCB
* Age ≥ 18 years
* Presence of a de novo lesion or in-stent restenosis in a native coronary artery or a in a bypass graft and suitable for PCI
* Reference vessel diameter between 2.0 - 4.5 mm
* Patient suitable for dual antiplatelet therapy (DAPT)

Exclusion Criteria:

* Inability to provide informed consent
* Allergy to paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) with stable CAD or ACS who have a PCI indication and are treated with the Protégé DCB.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
TLF at 1 year | From enrollment to 1 year follow-up
  Target Lesion Failure (TLF) at 1 year, defined as a composite of:
  * Cardiovascular death
  * Target vessel myocardial infarction (TV-MI)
  * Clinically driven target lesion revascularization (TLR)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands